CLINICAL TRIAL: NCT06374225
Title: Strategy to Avoid Excessive Oxygen Using an Autonomous Oxygen Titration Intervention (SAVE-O2 AI)
Brief Title: Strategy to Avoid Excessive Oxygen Using an Autonomous Oxygen Titration Intervention
Acronym: SAVE-O2 AI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); O2matic ApS (Unknown); IDTS Medical, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-0866
Record Dates: First submitted 2024-04-04; First posted 2024-04-18 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Critical Illness; Wounds and Injury; Disease Attributes; Pathologic Processes
Keywords: hypoxia; hyperoxia; burn; trauma; acute care surgery; acute respiratory illness; critical illness; supplemental oxygen; oxygenation; SpO2; PaO2; FiO2; normoxia; hypoxemia; hyperoxemia; normoxemia; autonomous; device
MeSH Terms: conditions — Critical Illness; Wounds and Injuries; Disease Attributes; Pathologic Processes; Hypoxia; Hyperoxia; Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Usual Care (Manual Titration) (No Intervention): Patients randomized to the usual care arm will receive usual care, manual oxygen titration, removal of supplemental oxygen, and escalation per hospital protocol, based on the site's usual SpO2 assessments. The SpO2 monitor for the O2matic PRO100 will also be connected to the patient in observation mode for data collection purposes only (not used for titration decisions).
- Intervention (Automated Titration) (Experimental): Patients randomized to the intervention arm will receive supplemental oxygen via nasal cannula (recommended up to 6 lpm) or face mask (recommended up to 15 lpm) and will have supplemental oxygen titrated using an autonomous oxygen titration system for the first 72 hours after randomization, or hospital discharge (whichever sooner).
  Interventions: Device: Automated Titration (O2matic)

INTERVENTIONS:
Device: Automated Titration (O2matic) — The patient will receive supplemental oxygen titrated using an autonomous oxygen titration device. The patient will be monitored and vital signs documented by the site's usual SpO2 assessments, but oxygen titration will occur automatically through the O2matic PRO100 device during the intervention period, unless there is a safety concern. The SpO2 range programmed into the PRO100 is 92-94%. The acceptable SpO2 range for the protocol is 90-96%. If a patient requires >15lpm or other signs of advancing respiratory failure, they will be taken off the autonomous oxygen and transitioned to higher flow oxygen devices or mechanical ventilation per usual clinical care. If the patient is not receiving any supplemental oxygen per the autonomous titration, the clinical team may remove the oxygen delivery device from the patient, but the patient should remain connected to the PRO100 for the duration of the intervention period for data collection and to monitor for new supplemental oxygen needs.
  Arms: Intervention (Automated Titration)

SUMMARY:
This study is a multicenter randomized controlled trial to determine the effectiveness of a closed loop/autonomous oxygen titration system (O2matic PRO100) to maintain normoxemia (goal range SpO2 90-96%, target 93%) during the first 72 hours of acute injury or illness, compared to standard provider-driven methods (manual titration with SpO2 target of 90-96%).

DETAILED DESCRIPTION:
Ensuring adequate oxygenation is a primary goal in surgical and medical patients to treat and prevent morbidity associated with hypoxemia. However, excessive oxygen administration resulting in hyperoxemia is common, leading to unnecessary utilization of supplemental oxygen, which is a particularly limited resource in austere settings. Building on the previous Strategy to Avoid Excessive Oxygen (SAVE-O2) clinical trials1 (Trauma: NCT045349559; Burn: NCT04534972), the investigators seek to determine effective strategies to implement a targeted normoxemia approach to avoid both hyperoxemia and hypoxemia and reduce supplemental oxygen use, using the PRO100 closed loop/autonomous oxygen system. This research is critical for both military and civilian care settings in determining the effectiveness of an autonomous oxygen system to use to 1) reduce harm associated with both hypoxemia and hyperoxemia and 2) reduce excess use of oxygen.

Objectives: the investigators propose the following two objectives:

Determine the effectiveness of an autonomous oxygen titration system to improve normoxemia and reduce hypoxemia and hyperoxemia in acutely injured and ill patients receiving supplemental oxygen. The investigators will compare patient-hours spent in normoxemia (SpO2 90-96%), hypoxemia (SpO2 <88%), and hyperoxemia (SpO2 >96%) among patients randomized to autonomous vs manual oxygen titration.

Determine the impact of an autonomous oxygen titration system on overall utilization of supplemental oxygen. The investigators will compare the total volume of supplemental oxygen administered to patients randomized to autonomous vs manual oxygen titration during the 72-hour intervention period.

Hypothesis: The investigators hypothesize that the use of an autonomous oxygen titration system will be more effective at maintaining normoxemia and reducing time spent in hypoxemia/hyperoxemia than standard manual titration in non-mechanically ventilated patients and will reduce the overall use of supplemental oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Hospitalized or will be hospitalized from Emergency Department for major trauma, burn, acute care surgery, or acute respiratory illness
* Able to be randomized within 36 hours of hospital arrival
* Receiving supplemental oxygen 1-10 liters per minute for documented or presumed hypoxemia (must be higher than baseline for those on chronic oxygen therapy)
* Signed and dated informed consent from patient or legally authorized representative (LAR)

Exclusion Criteria:

* Anticipated hospital discharge within 24 hours
* Imminent plans to discontinue supplemental oxygen
* Imminent plans to administer high flow nasal oxygen, non-invasive ventilation, or invasive mechanical ventilation
* Clinical team unwilling or unable to follow the prescribed oxygen titration method in either randomized group
* Known prisoner
* Known pregnancy
* Known contraindicated conditions for use of the PRO100 device: carbon monoxide poisoning, incapable of handling airway secretions, increased methemoglobin, cyanide poisoning, cluster headaches, undrained pneumothorax, sickle cell crisis, paraquat poisoning or a history of bleomycin poisoning, patients for whom the SpO2 signal is not stable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-12-07 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of time spent within the targeted normoxemia range | during first 72 hours after randomization, censored at hospital discharge, escalation to high flow nasal oxygen/mechanical ventilation, or death if prior to 72 hours.
  The primary endpoint is proportion of time spent within the targeted normoxemia range, defined as an oxygen saturation (SpO2) of 90-96% (target 93%), as measured by continuous non-invasive pulse oximetry, during the first 72 hours after randomization, censored at hospital discharge, escalation to high flow nasal oxygen/mechanical ventilation, or death if prior to 72 hours.

SECONDARY OUTCOMES:
Amount of supplemental oxygen administered | during first 72 hours after randomization
  defined as total estimated oxygen volume during the first 72 hours after randomization.
Proportion of time spent in hypoxemia (SpO2<88%) | during first 72 hours after randomization
  Proportion of time spent in hypoxemia (SpO2 <88%) during the first 72 hours after randomization.
Proportion of time spent in hyperoxemia (SpO2 >96%) | during first 72 hours after randomization
  Proportion of time spent in hyperoxemia (SpO2 >96%) during the first 72 hours after randomization.
Time to Room Air | censored at day 28, discharge if before day 28, or death.
  defined as the time from hospital presentation to the first episode of no supplemental oxygen (room air), censored at discharge or death.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Colorado, Aurora, Colorado
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Oregon Health and Sciences University, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Douin DJ, Rice JD, Xiao M, Beaty L, Guo C, Withers C, Sullivan A, Anderson EL, Cheng AC, Banasiewicz MK, Semler MW, Lloyd BD, Maiga A, Gibbs KW, Stettler GR, Khan A, Sally MB, Wright FL, Aggarwal N, Bebarta VS, Ginde AA; SAVE-O2 AI Investigators. Statistical analysis plan for the Strategy to Avoid Excessive Oxygen using Autonomous Oxygen Titration Intervention (SAVE-O2 AI) trial: protocol. BMJ Open. 2026 Jan 28;16(1):e110739. doi: 10.1136/bmjopen-2025-110739. PMID 41605593